CLINICAL TRIAL: NCT02307669
Title: A Study on Inhaler Adherence to Improve Poor Asthma Control
Brief Title: Inhaler Adherence in Severe Unstable Asthma
Acronym: INCA-SUN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Professor Richard Costello, Professor of Medicine, Beaumont Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: INCA-Sun
Record Dates: First submitted 2014-04-21; First posted 2014-12-04 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Asthma
Keywords: Adherence; Inhaler; GINA
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Routine inhaler adherence care (Placebo Comparator): Normal Care group This management is based on the inhaler training recommendations of the BTS/SIGN group (http://www.brit-thoracic.org.uk/Portals/0/Guidelines/AsthmaGuidelines/sign101%20Jan%202012.pdf) and medication management of the GINA management strategy.
  The core features of the "usual care" group are:
  1. The patient's inhaler technique will be checked using a checklist, at each visit. If there are errors these will be corrected using teach-to-goal principals.
  2. Adherence will be discussed and barriers to adherence addressed, using motivational interview techniques.
  3. Written action plans for managing asthma, based on changes in PEF and symptoms will be given.
  4. In follow up, medication changes in response to the above will be directed by these, as suggested by GINA management guidelines using a standardised digital script.
  Interventions: Behavioral: Usual Care
- INCA feedback (Active Comparator): 1. The patient's treatment goal is established and used as the focus of the conversation.
  2. Data from the INCA device including (1) time of use, (2) handling proficiency and (3) inhalation flow rates are discussed, with three graphs as shown in the appendix and derived as discussed. These are aimed to enhance the value of the inhaler.
  3. Data from the electronic PEF and AQLQ are correlated with digitally recorded adherence so that these can be used to account for improvements or declines in these measures.
  4. In follow up, medication changes in response to the above (adherence, PEF, ACT and exacerbations) are made using a standardised digital script.
  Interventions: Behavioral: INCA feedback

INTERVENTIONS:
Behavioral: INCA feedback — The study team have developed a device which is attached to inhalers that makes an audio recording of the inhaler being used. Analysis of this audio data provides objective evidence of the time of inhaler use, technique of use and the peak inspiratory flow the patient makes each time they use their inhaler. Our preliminary experiences with the information obtained from this device indicate that adherence is poor in patients with severe asthma due to any one the following issues poor time of use, errors in handling and low peak inspiratory flow rates.
  Arms: INCA feedback
Behavioral: Usual Care — The core features of the "usual care" group are:
  The patient's inhaler technique will be checked using a checklist, at each visit. If there are errors these will be corrected using teach-to-goal principals.
  Adherence will be discussed and barriers to adherence addressed, using motivational interview techniques.
  Written action plans for managing asthma, based on changes in PEF and symptoms will be given.
  In follow up, medication changes in response to the above will be directed by these, as suggested by Guidelines.
  Arms: Routine inhaler adherence care

SUMMARY:
The investigators hypothesize that aligning digital data on PEF and adherence with the patient's own clinical course achieves better asthma control and identifies risks for future loss of control, compared to current best practice. The study has an adherence optimisation phase, week 1-12 followed by a medication management phase, week 12 to week 32.

The investigators will compare two asthma education interventions, standard Guideline recommended practice and feedback from the individual's own INCA device, which assesses inhaler adherence and relates adherence with changes in PEF and symptom scores over time.

The study has two co-primary endpoints, one will be a comparison of the adherence to therapy and the other will be a comparison of the appropriateness of medication prescriptions between the two study groups.

DETAILED DESCRIPTION:
The investigators hypothesize that aligning adherence, inhaler technique and digitally recorded PEF to inform patients and as the basis of prescribing decisions achieves better inhaler adherence and technique and also allows physicians to make appropriate prescribing decisions, compared to current best practice.

The investigators will compare two asthma education interventions, standard BTS/SIGN Guideline recommended practice and feedback from the individual's own INCA device, which assesses inhaler adherence and relates adherence with changes in PEF and symptom scores over time.

This education phase is followed by a medication optimisation phase (weeks 12-32) in which there are 3 cycles of medication optimisation guided by a digital script. The script either adjusts the medications following the GINA recommendation or uses the GINA recommendation but is supplemented with data on adherence and PEF that are recorded to digital, time-stamped, recording devices.

The aim of the study is to improve and maintain adherence to preventer therapy, so that medication and other costs as well as the quality of life, exacerbation rates are optimal.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to give voluntary informed consent
* Must have a clinical diagnosis of asthma supported by objective measures, one of the following by FEV1/FVC <70% and FEV1 <80% or - a 12% change in FEV1 following administration of a beta-agonist or spontaneously over 1 year period, a positive bronchial provocation test, or a 10% variability in PEF within a 7 day period.
* Must have a bronchodilator FEV1 > 40% and <80% in the past 1 year
* Current unstable asthma i.e. ACT score ≤ 19 at enrolment despite already being managed with GINA step 3-5 therapy.
* One or more courses of oral corticosteroids in the prior year, or a hospitalization or ED attendance with an asthma exacerbation in the last year
* Age 18 years or older at time of consent.
* Capable of understanding and complying with the requirements of the protocol, including the ability to attend for all required visits.
* Able and willing to take inhaled medication via a Diskus.
* In the opinion of the investigator suitable for use of a salmeterol/fluticasone Diskus inhaler or already using a salmeterol/fluticasone inhaler.

Exclusion Criteria:

* Have used any investigational product or device within 3 months of the enrolment visit.
* Have known previous sensitivity to Seretide (salmeterol/fluticasone).
* Have a known significant (in the opinion of the investigator) concurrent medical disease, pregnancy that might mean that the participant cannot complete the study.
* Be taking omalizumab or other biological agent used in the treatment of asthma
* Concurrent treatment with potent cytochrome P450 3A4 (CYP3A4) inhibitors; Ketoconazole and Ritonavir.

  * Current smokers and ex-smokers with a greater than 20 pack year history of cigarette smoke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-01-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean rate of actual Adherence to preventer medication | week 20 through 32
  This study will focus on severe asthma patients, who remain uncontrolled and with frequent exacerbations requiring oral steroids and have an Asthma control test (ACT) score of <19 on enrollment.
The between-group difference in the proportion of patients prescribed guideline appropriate medication at the end of the study. | week 20 through 32
  The appropriateness of the prescribed therapy will be verified for each participant after study completion using all available adherence and PEF data.
  Between-group differences will be further broken down by the following:
  * The proportion of participants prescribed add-on therapy (e.g. Monoclonal antibody therapy)
  * The proportion of participants whose ICS/LABA dose was increased
  * The proportion of participants whose ICS/LABA dose was reduced

SECONDARY OUTCOMES:
Cost-effectiveness and economic evaluation of the INCA educational intervention | First 8 weeks of the study and week 20 to 32
  An economic evaluation of national implementation of the INCA-SUN program will be provided. Data on the cost of the intervention (device, time taken to deliver, cost of training and salary cost of the trainer), medication costs, quality of life, exacerbations and other healthcare utilization and associated costs, such as unscheduled health care visits as well as work productivity losses will be collected alongside the 32-week study.
  A cost-effectiveness and cost-utility analysis of the intervention compared to the control arm will be performed. Incremental cost-effectiveness ratios (or ICERS) will be calculated from the data, to estimate how much additional cost is required for an additional unit of benefit.
Change in Asthma Control Test scores at week 32 | Baseline to week 32
  ACT scores will be obtained during the study visits.
Change in PEF variability | Baseline to week 32
  Differences between the two study groups will be calculated
Change in AQLQ | Baseline to week 32
  AQLQ scores will be obtained during the study visits.
Exacerbations over study period | Baseline to week 32
  It is hypothesised that with active education, exacerbation frequency can be reduced.
To compare the proportion of patients who were clinically stable | First 8 weeks of the study and week 20 to 32
  The proportion of patients who required no daily reliever use in the month prior to study end will be compared.
Relationship of biomarkers with adherence | Baseline to week 32
  A comparison of changes in blood eosinophil's, periostin and Fractional Exhaled Nitric Oxide (FeNO) between the active and control groups will be made.The relationship between 7-day FeNO suppression and clinical and biomarker outcomes will be investigated.10. The relationship between changes in FeNO (characterised into FeNo>45ppb Or FeNO<45ppb) and adherence will also be investigated.
The proportion of patients who are refractory to treatment | First 8 weeks of the study and week 20 to 32
  A comparison of the proportion of patients who are refractory, (defined as having actual adherence ≥80%, ≥1 exacerbation, PEF am/pm <80% and ACT ≤19) will be conducted.
The proportion of patients who are non-adherent and remain uncontrolled | First 8 weeks of the study and week 20 to 32
  The proportion of patients who are non-adherent and remain uncontrolled, (i.e. Actual Adherence <80%, PEF am/pm <80% and ACT≤19) between the active and control groups will be compared.
The proportion of patients with inhaler related side effects | First 8 weeks of the study and week 20 to 32
  The proportion of patients with inhaler related side effects including oral candidiasis between the active and control groups will be compared.

OTHER OUTCOMES:
Patient identified goal | Baseline to week 32
  Proportion of patients reaching stated clinical goal at week 12 and between that period and week 32.

CONTACTS AND LOCATIONS:
Overall Officials: Richard w Costello, MD, Principal Investigator — RCSI
Locations (1):
- Beaumont Hospital, Dublin, Ireland

REFERENCES:
- [Background] Mokoka MC, Lombard L, MacHale EM, Walsh J, Cushen B, Sulaiman I, Carthy DM, Boland F, Doyle F, Hunt E, Murphy DM, Faul J, Butler M, Hetherington K, Mark FitzGerald J, Boven JFV, Heaney LG, Reilly RB, Costello RW. In patients with severe uncontrolled asthma, does knowledge of adherence and inhaler technique using electronic monitoring improve clinical decision making? A protocol for a randomised controlled trial. BMJ Open. 2017 Jun 15;7(6):e015367. doi: 10.1136/bmjopen-2016-015367. PMID 28619778
- [Derived] Hale EM, Greene G, Mulvey C, Mokoka MC, van Boven JFM, Cushen B, Sulaiman I, Brennan V, Lombard L, Walsh J, Plunkett S, McCartan TA, Kerr PJ, Reilly RB, Hughes C, Kent BD, Jackson DJ, Butler M, Counihan I, Hayes J, Faul J, Kelly M, Convery R, Nanzer AM, Fitzgerald JM, Murphy DM, Heaney LG, Costello RW; INCA Research Team. Use of digital measurement of medication adherence and lung function to guide the management of uncontrolled asthma (INCA Sun): a multicentre, single-blinded, randomised clinical trial. Lancet Respir Med. 2023 Jul;11(7):591-601. doi: 10.1016/S2213-2600(22)00534-3. Epub 2023 Mar 21. PMID 36963417
- [Derived] Butler CA, Heaney LG. Fractional exhaled nitric oxide and asthma treatment adherence. Curr Opin Allergy Clin Immunol. 2021 Feb 1;21(1):59-64. doi: 10.1097/ACI.0000000000000704. PMID 33369570

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT02307669/SAP_000.pdf